CLINICAL TRIAL: NCT06826664
Title: Creation, Management and Analysis of a National Database of Patients Affected by Diseases of Phosphate Metabolism
Brief Title: Institution of an Italian Multicenter Database of Patients Affected by Diseases of Phosphate Metabolism
Status: Not yet recruiting | Type: Observational
Sponsor: F.I.R.M.O. - Fondazione Italiana Ricerca sulle Malattie dell'Osso - Ente del Terzo Settore (Other)
Responsible Party: Sponsor
Other Study IDs: 24033_oss
Record Dates: First submitted 2025-01-22; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Phosphate Deficiency; Phosphate Overload
Keywords: Phosphate; Phosphate metabolism; Hyperphosphatemia; Hypophosphatemia; Retro-prospective clinical data collection; Database of patients
MeSH Terms: conditions — Hyperphosphatemia; Hypophosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected by diseases of phosphate metabolism: A single cohort of male and female patients of any age who are affected by one disease of phosphate metabolism.
  The observational study does not include any type of intervention.

SUMMARY:
The goal of this observational study is to create, manage and analyze a multicenter national database of patients affected by diseases of phosphate metabolism, aimed at collecting and studying anamnestic, diagnostic, genetic, clinical, and therapeutic data in a relatively wide number of patients with these rare inherited metabolic disorders in Italy.

The study will include 28 specialist clinical centers of endocrinology, pediatric endocrinology, and pediatrics, located throughout the Italian territory, and to which patients refer from all the 20 regions of Italy.

Data will be collected over time, both in retrospective and prospective manners, during the 10-year duration of the study, starting from the recruiting visit (basal visit) and then during each follow-up visits patients will undergo for the control of disease at the recruiting clinical centers.

Collected data will include both the most classic traits of each disease and the less common ones, with the final goal of refining and deepening medical knowledge in the field of these rare inherited metabolic disorders, and, thus, to be able to define optimal tailored diagnostic, clinical, and therapeutic management of patients, improving their quality of life.

The main aspects this observational study aims to assess and clarify are:

1. Evaluation of prevalence and incidence of diseases of phosphate metabolism in Italy, globally and for single different disorders
2. Clinical and biochemical characterization of different diseases of phosphate metabolism (according to single disorders and different genetic base), through both cross-sectional and longitudinal analyses of collected data
3. Evaluation of skeletal health and bone fragility in patients with diseases of phosphate metabolism, globally and based on single phosphate metabolism disorder, gender, and age
4. Self-evaluation of health-related quality of life in patients with a disease of phosphate metabolism
5. Over time evaluation of responses to therapies in patients with diseases of phosphate metabolism.

The study will include a single cohort of female and male patients of any age, affected by a disease of phosphate metabolism. The study does not include either any control group/comparison group or healthy volunteers.

The study itself does not involve any medical intervention or drug administration. Therapies for which response outcomes will be collected in the database, are those commonly employed for the treatment of diseases of phosphate metabolism, regardless of patients' inclusion in this observational study.

DETAILED DESCRIPTION:
1. Background and rationale

   Phosphorus is one of the most abundant elements in the human body, where it is found, mainly in the form of phosphate salts, in quantities of about 500-700 grams, of which about 85% is concentrated in bone tissue, where it is an important constituent of hydroxyapatite crystals. In soft tissues, phosphate is mainly found in the intracellular compartment as an essential component of various organic compounds, including nucleic acids and phospholipids of the cell membrane.

   The concentration of circulating extracellular phosphate is finely regulated by hormones such as parathyroid hormone (PTH), the active form of vitamin D (1,25-dihydroxyvitamin D or calcitriol), and fibroblast growth factor 23 (FGF23). The latter belongs to a family of proteins, specifically responsible for regulating phosphate metabolism, which are called phosphatonins in their complex, and include FGF23, Phosphate Regulating Endopeptidase X-Linked (PHEX), Polypeptide N-Acetylgalactosaminyltransferase 3 (GALNT3), Klotho. Under normal conditions, the coordinated action of phosphotropic hormones modulates intestinal absorption of this mineral, its renal reabsorption, and bone mineralization, maintaining the balance between absorption and excretion and ensuring a normal blood concentration of phosphate between 2.5 and 4.5 mg/dl (0.81-1.45 mmol/L) in the adult organism. Bone phosphate serves as a deposit, capable of buffering changes in plasma and intracellular levels of phosphate. Alterations in the mechanisms that regulate phosphate metabolism are responsible for the development of a group of rare disorders that are collectively defined as phosphate metabolism diseases, and include diseases caused by excess phosphate (hyperphosphatemic disorders), such as calcinosis, and diseases caused by deficiency of phosphate (hypophosphatemic disorders), such as hypophosphatemic rickets.

   Phosphate metabolism diseases are classified as rare diseases. As reported by the "Osservatorio Malattie Rare (OMAR)", in the European Union a disease is defined as rare when its prevalence, understood as the number of cases present in a given population, is less than 0.05 percent of the population (no more than one case in every 2,000 people). The rarity of these diseases makes them difficult to study, and unfortunately, in many cases, scientific and medical knowledge of rare diseases is scarce and inadequate, and limited to few case reports. Due to the lack of sufficient medical and scientific knowledge, many patients affected by rare diseases remain undiagnosed and their diseases remain unrecognized. It is, therefore, essential that doctors and researchers working in the field of rare diseases increasingly work in networks to share the results of their research and to progress more effectively in the knowledge and clinical management of these diseases. In this perspective, implementing and detailing as much as possible the knowledge on the epidemiology, clinical and therapeutic history, primary and secondary manifestations of diseases of phosphate metabolism and the response to employed therapies, both in cross-sectional and longitudinal manners, with constant follow-up assessments of patients is essential not only to improve the clinical management of single patients, but also to allow better planning of social, political and health interventions for these pathologies and, overall, improve the quality of life of patients.

   For this reason, it is extremely important to create a national multicenter database, such as the one proposed by this study, which is able to collect a relatively high number of patients affected by diseases of phosphate metabolism, whose cases are carefully studied in every aspect, both retrospectively and prospectively, following the course of the disease over time. Such a database has never been prepared in Italy before, and the availability of clinical data relating to diseases of phosphate metabolism has been limited to individual clinical cases to date.

   The collection of clinical data of patients affected by diseases of phosphate metabolism, both retrospectively (during the study recruitment visit) and prospectively (during follow-up visits), will allow for an epidemiological evaluation of these pathologies in Italy and for both cross-sectional and longitudinal analyses of the collected data, with particular attention to the clinical evolution, response to therapies, and quality of life of the patients.
2. Main aim and specific objectives

Main goal of this observational study is to create, manage and analyze a retro-prospective multicenter national database of patients affected by diseases of phosphate metabolism, aimed at collecting and studying anamnestic, diagnostic, genetic, clinical, and therapeutic data in a relatively wide number of patients with these rare congenital metabolic disorders in Italy.

Such a database will allow for an epidemiological evaluation of prevalence and incidence of diseases of phosphate metabolism in Italy, and to collect case history of patients whose clinical cases will be studied in detail and followed over time up to 10 years after the recruitment in the study, in order to refine knowledge in the field of these rare disorders.

Specific objectives of the studies are:

1. Creation of an Italian centralized multicenter database of patients affected by diseases of phosphate metabolism, through the collection of patients at 28 specialist clinical centers of endocrinology, pediatric endocrinology, and pediatrics, located throughout the Italian territory and visiting patients from all the 20 regions of Italy.
2. Collection of a relatively high number of patients affected by diseases of phosphate metabolism
3. Retrospective collection of data about diseases of phosphate metabolism, at the time of the recruiting visit.
4. Continuous and updated prospective collection of patients' data over time, starting from the first recruiting visit up to 10 years after the recruitment in the study.

6. Evaluation of prevalence and incidence of diseases of phosphate metabolism in Italy, globally and for single different disorders 7. Clinical and biochemical characterization of different diseases of phosphate metabolism (according to single disorders and different genetic base), through both cross-sectional and longitudinal analyses of collected data 8. Evaluation of skeletal health and bone fragility in patients with diseases of phosphate metabolism, globally and based on single phosphate metabolism disorder, gender, and age 9. Self-evaluation of how the disease of phosphate metabolism interferes on the quality of life, daily activities, work, and emotional state of affected patients 10. Over time evaluation of responses to therapies in patients with diseases of phosphate metabolism.

3. Study population

The study will include a single cohort of female and male patients of any age, affected by a disease of phosphate metabolism.

The study does not include either any control group/comparison group or healthy volunteers.

Diseases of phosphate metabolism are classified as rare diseases and there are no data available on their true prevalence, as a whole. The prevalence of some specific phosphate metabolism disorders, such as X-linked hypophosphatemia (1-9/100,000), autosomal dominant hypophosphatemic rickets (< 1/1,000,000), dominant hypophosphatemia with nephrolithiasis or osteoporosis (< 1/1,000,000), is available on the Portal for Rare Diseases and Orphan Drugs (Orphanet). Based on the prevalence data available those single phosphate metabolism disorders on Orphanet we can estimate that a minimum of 100 patients will be globally collected in the present study.

3.1 Inclusion criteria

* Clinical and/or genetic diagnosis of a rare disease of phosphate metabolism 3.2 Exclusion criteria
* None

  4. Study design and setting

Non-profit, multicenter, national, retro-prospective, observational study, consisting in the design, creation, management and analysis of an Italian database of patients affected by diseases of phosphate metabolism.

The study will last 10 years. The enrollment of patients, the inclusion in the database with retrospective collection of their clinical data, and the subsequent prospective collection of clinical follow-up data will take place throughout the duration of the study. For the retrospective collection, retrospective data on the disease of phosphate metabolism will be retrieved from patient's medical records, at the time of the medical visit that the patient will carry out at the Clinical Center for the evaluation of his/her disease, regardless of inclusion in this study. Prospective data relating to the follow-up of disease of phosphate metabolism will be collected during the subsequent medical follow-up visits, scheduled for each patient as part of the clinical management of his/her clinical condition, regardless of inclusion in this study.

Being an observational study, this study itself does not involve the administration of any drug, nor the use of any medical device, nor does it involve additional medical visits, clinical analyses or care procedures in addition to those conventionally scheduled for the clinical and therapeutic management of patient affected by a disease of phosphate metabolism. No participant biospecimens of any type will be collected and retained to perform this study. Therapies for which data on response outcomes will be collected in the database, are those usually employed for the treatment of patients with diseases of phosphate metabolism, regardless of their inclusion in this observational study.

All data will be collected anonymously, and they will be analyzed as aggregates. Data collected in the database will be, first, processed using descriptive statistics, such as frequency tables for categorical data, median and quartiles for quantitative data on ordinal scales and mean and standard deviation for quantitative data on metric scales. Secondly, the correlations between variables will be evaluated using the Pearson correlation index in the case of continuous variables and the chi-square test for categorical variables.

5. Data and variables

Data collected in the database will include (if available in patient's medical records and part of the normal clinical and therapeutic management of patient regardless of inclusion in this study):

* Demographics (sex, year of birth)
* Age at diagnosis/onset of disease of phosphate metabolism
* Personal clinical history of disease of phosphate metabolism
* Family history of disease of phosphate metabolism in first-degree relatives
* Presence of comorbidities
* Result of the genetic testing for genes known to be involved in the development of congenital diseases of phosphate metabolism
* Clinical manifestations of the disease and related signs and symptoms
* Over time evaluation of biochemical parameters of metabolism of phosphate (i.e phosphatemia and 24h phosphaturia)
* Over time biochemical evaluation of kidney function (i.e. creatinine, clearance of creatinine, estimated glomerular filtration rate, spot proteinuria, 24h proteinuria)
* History of fragility fractures, bone deformities and altered musculoskeletal development
* Over time evaluation of biochemical parameters of calcium and bone metabolism (i.e calcemia, calcium ion, 24h calciuria, 25(OH)-vitamin D, 1,25(OH)2-vitamin D, parathyroid hormone, bone alkaline phosphatase, serum carboxy-terminal collagen crosslinks, serum procollagen 1 N-terminal propeptide)
* Over time skeletal X-ray analysis (absence/presence of vertebral fracture, osteomalacia, of calcinosis, not healing fractures, extra skeletal calcifications)
* Over time instrumental assessment of bone mineral density and bone tissue microstructure [assessed by Dual-energy X-ray absorptiometry (DXA), Radiofrequency Echographic Multi Spectrometry (REMS), peripheral Quantitative Computed Tomography (pQCT), and/or High-Resolution pQCT (HR-pQCT)]
* Self-evaluation of health-related quality of life through the 36-Item Short Form Health Survey (SF-36) questionnaire
* Pharmacological therapies (drug, duration, posology)
* Disease-related morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* Clinical and/or genetic diagnosis of a rare disease of phosphate metabolism

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A single cohort of female and male patients of any age, affected by a disease of phosphate metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2035-05-31 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence and incidence evaluation | Through study completion, an average of 10 years
  Evaluation of prevalence and incidence of diseases of phosphate metabolism, globally and for single different disorders
Clinical characterization of diseases of phosphate metabolism | Through study completion, an average of 10 years
  Detailed clinical characterization of each different rare disease of phosphate metabolism performed through retrospective and prospective cross-sectional and longitudinal collection of available data on disease clinical history, over time clinical manifestations and their age of onset, and related signs and symptoms.
  For each disease, the collected clinical features will be analyzed through descriptive statistical analyses and expressed as percentage of frequency for categorial data and as mean/median value for continuous data.
Biochemical parameters of phosphate metabolism | Through study completion, an average of 10 years
  Over time assessment of metabolism of phosphate, in each different rare disease, through the collection of data on specific biochemical parameters, at baseline visit and during follow-ups:
  * Serum phosphate (mg/dl)
  * 24h phosphaturia (mg/24h) Each biochemical parameter will be, singularly, categorized as reduced levels, normal levels, or increased levels, according to its reference values, and analyzed through descriptive statistical analyses as percentage of frequency.
Biochemical parameters of kidney function | Through study completion, an average of 10 years
  Over time assessment of kidney function, in each different rare disease of phosphate metabolism, through the collection of data on specific urinary parameters, at baseline visit and during follow-ups:
  * Creatinine (mg/dl)
  * Clearance of creatinine (ml/min)
  * Estimated Glomerular Filtration Rate (eGFR) (mL/min/1.73 m2)
  * Spot proteinuria (mg/dl)
  * 24h proteinuria (mg/24h) Each biochemical parameter will be, singularly, categorized as reduced levels, normal levels, or increased levels, according to its reference values, and analyzed through descriptive statistical analyses as percentage of frequency.
Descriptive analyses of skeletal health and bone fragility in patients with diseases of phosphate metabolism | Through study completion, an average of 10 years
  Over time assessment of skeletal health and bone fragility:
  1. History of fractures, bone deformities, altered musculoskeletal development
  2. Calcium and bone metabolism:
     Calcemia (mg/dl) Calcium ion (mg/dl) 24h calciuria (mg/24h) Parathyroid hormone (pg/ml) 25(OH)-vitamin D (ng/ml) 1,25(OH)2-vitamin D (pg/ml) Bone alkaline phosphatase (mcg/L) Serum carboxy-terminal collagen crosslinks (CTX) (ng/ml) Serum procollagen 1 N-terminal propeptide (P1NP) (ng/ml)
  3. Skeleton X-ray: presence/absence of vertebral fracture, osteomalacia, calcinosis, not healing fractures, extra skeletal calcifications
  4. Instrumental bone evaluation: bone mineral density (g/cm2), T-scores, Z-scores Biochemical parameters will be categorized as reduced, normal, or increased levels, according to their reference values For each disease, data will be singularly analyzed by descriptive statistical analyses, and expressed as percentage of frequency for categorial data and as mean/median value for continuous data
Assessment of health-related quality of life in patients with a disease of phosphate metabolism | Through study completion, an average of 10 years
  Self-evaluation of how the disease interferes with quality of life, daily activities, work, and emotional state of the affected patient, through the Short Form Health Survey 36 (SF-36) questionnaire.
  The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Component analyses measure two distinct concepts: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).
Assessment of response to targeted therapy in patients with diseases of phosphate metabolism | Through study completion, an average of 10 years
  Over time evaluation of the response to therapy in patients with a specific disease of phosphate metabolism for which a targeted therapy for that disease is approved, and who are under treatment independently by the participation to this observational study.
  Rate of efficacy of each treatment will be assessed among treated patients, by evaluating how medication is able to: 1) control/restore the correct phosphate metabolism over time, 2) alleviate, reduce or eliminate signs and symptoms of the disease, 3) prevent disease progression and/or worsening, 4) ameliorate the quality of life of patient.
  Side effects and adverse events directly related to each drug, and reported in patient's clinical record, will be evaluated, each, as percentage of frequency.

CONTACTS AND LOCATIONS:
Locations (28):
- Italy (28):
  - U.O.C. Endocrinologia, Azienda Ospedaliero Universitaria Policlinico Consorziale, Università degli Studi di Bari "Aldo Moro", Bari
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, UO Pediatria, Programma di Malattie Endocrino-Metaboliche, Bologna
  - UOC Endocrinologia e Prevenzione e Cura del Diabete, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Dipartimento di Scienze Mediche e Chirurgiche (DIMEC), Alma Mater Studiorum Università di Bologna, Bologna
  - Centro di Auxoendocrinologia e Genetica Medica della Clinica Pediatrica degli Spedali Civili di Brescia, Brescia
  - Endocrinologia e Diabetologia, Azienda Ospedaliero-Universitaria di Cagliari, Presidio Ospedaliero Policlinico di Monserrato, Cagliari
  - UO Endocrinologia e Malattie del Ricambio, Azienda Ospedaliero Universitaria di Ferrara, Sezione di Endocrinologia, Geriatria e Medicina Interna, Dipartimento di Scienze Mediche, Università degli Studi di Ferrara, Ferrara
  - Diabetologia e Endocrinologia, Auxoendocrinologia, Children's Hospital Meyer IRCCS, Florence
  - SOD Malattie del Metabolismo Minerale ed Osseo, Azienda Ospedaliero-Universitaria Careggi, Florence
  - Clinica Endocrinologica, Dipartimento di Medicina Interna e Specialità Mediche (DiMI), IRCCS Ospedale Policlinico San Martino, Università di Genova, Genova
  - Clinica Pediatrica ed Endocrinologia, IRCCS Ospedale Pediatrico Giannina Gaslini, Genova
  - Dipartimento di Patologia Umana dell'adulto e dell'età evolutiva "Gaetano Barresi", Università degli Studi di Messina, Messina
  - UOC di Endocrinologia, AOU Policlinico G. Martino, Dipartimento di Patologia Umana DETEV, Università di Messina, Messina
  - Dipartimento di Malattie Endocrino-Metaboliche, IRCCS Istituto Auxologico Italiano, Milan
  - Dipartimento di Pediatria, IRCCS Ospedale San Raffaele, Milan
  - SC Endocrinologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Dipartimento di Pediatria, Azienda Universitaria Ospedaliera della Seconda Università degli Studi di Napoli, Napoli
  - Clinica Medica 1, Dipartimento di Medicina, Università di Padova, Padua
  - UOC Endocrinologia, DIMED, Azienda Ospedaliero-Universitaria di Padova, Padua
  - Centro di Riferimento Regionale Toscano per l'Endocrinologia Pediatrica, Azienda Ospedaliero Universitaria Pisana, Pisa
  - Unità Operativa Endocrinologia 2, Azienda Ospedaliera Universitaria Pisana, Pisa
  - Unità di Endocrinologia e Andrologia, Dipartimento di Medicina Clinica e Molecolare, AOU Sant'Andrea, Centro di eccellenza ENETS, Università Sapienza di Roma, Roma
  - UOC di Endocrinologia e Diabetologia, UOS di Endocrinologia Pediatrica, IRCCS Ospedale Pediatrico Bambino Gesù, Roma
  - Donatello Bone Clinic, Casa di Cura Villa Donatello, Sesto Fiorentino
  - Endocrinologia Pediatrica Ospedale Infantile regina Margherita-Dipartimento di Scienze di Sanità Pubblica e Pediatriche, Università degli studi di Torino, Torino
  - SCDU Endocrinologia Diabetologia e Malattie del Metabolismo, AOU Città della Salute e della Scienza di Torino, Università di Torino, Torino
  - IRCCS Materno-Infantile Burlo Garofolo, Trieste
  - SOC Endocrinologia, Azienda Sanitaria-Universitaria Friuli Centrale, Udine
  - Unità di Reumatologia, Dipartimento di Medicina, Università di Verona, Verona